CLINICAL TRIAL: NCT05790343
Title: Feasibility Study of Empowering Parents Empowering Communities: Being a Parent Helping Your Child With Fears and Worries (BAPHYC)
Brief Title: Feasibility Study: Being a Parent - Helping Your Child With Fears and Worries
Acronym: BAPHYC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: King's College London (Other)
Collaborators: University of Oxford (Other); South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: BAPHYC - April 2022 V1.0
Record Dates: First submitted 2023-03-02; First posted 2023-03-30 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-01

CONDITIONS: Feasibility; Anxiety; Empowerment; Peer Influence
Keywords: Peer led intervention
MeSH Terms: conditions — Anxiety Disorders; Empowerment

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BAPHYC: Parents of children, aged 5-12 years, who have anxiety problems.
  Interventions: Behavioral: BAPHYC

INTERVENTIONS:
Behavioral: BAPHYC — Nine weekly peer led group meetings

SUMMARY:
Emotional disorders are among the most common childhood mental health difficulties. The majority of adult emotional disorders begin before age 14 years. Most children and families across the population do not receive the proven evidence-based interventions available, particularly those from socially disadvantaged neighbourhoods and excluded, Black and Minoritised populations. Families from disadvantaged neighbourhoods, Black and minoritised communities can often feel judged, mistrustful, and blamed for their children's behavioural difficulties making them reluctant to engage in parenting supportEven when available, research shows that over one-third of parents receiving traditional specialist delivered evidence-based parenting do not gain the expected outcomes. Undertaking a group-based parenting intervention to help parents understand and deal with their children's anxiety issues. The aim of this study is to examine the feasibility and acceptability of a new parent-led parenting intervention, being a Parent Helping your Child (BAPHYC) that is intended to improve childhood anxiety and to use the findings to inform the planning and conduct of a definitive randomised control trial.

Being a Parent- Helping your Child (BAPHYC) has been developed from two well-established evidence-based parenting programmes. It is a parent-led, group format manualised parenting programme intended to improve childhood anxiety in children aged 5-12 years consisting of eight two-hourly weekly sessions peer-facilitated by two trained parent group leaders. The particants of BAPHYC participants are mothers, fathers and other carers who have principal parenting responsibility for a child with anxiety.

The specific study objectives are to:

1. Establish initial evidence about reach and engagement, delivery, acceptability and impact of BAPHYC
2. Establish the feasibility of proposed recruitment pathways and measure completion
3. Acquire a fine grain understanding of parents' experiences of the BAPHYC intervention, research procedures and themes arising from BAPHYC implementation.
4. Assess participant recruitment, engagement, intervention and measure completion, and intervention acceptability rates against a priori feasibility parameters.
5. Obtain data that will be used in future trial recruitment and planning.

DETAILED DESCRIPTION:
Peer-led intervention models are a promising method for providing effective and acceptable parenting support to families considered hard to reach by mainstream services. Empowering Parents, Empowering Communities (EPEC) is an established parenting programme that involves recruiting and training local parents as "peer facilitators" to deliver manualised, evidence-based parent training groups in socially disadvantaged communities. EPEC optimises existing skills and relationship within local socially disadvantaged communities to deliver high quality, evidence-based parenting support for hard-to-reach families. Its group-based parenting course format is consistent with policy recommendations and intended to build social support between participants, optimise impact, and lower unit cost. EPEC is delivered in local, community locations and uses high visibility, pro-active local outreach campaigns to engage parents. Within these targeted community locations, an open access approach is typically used, rather than formal referral. To date, EPEC has focussed on increased scale of community-based care from birth to adolescence particularly in relation to behavioural and neurodevelopmental difficulties. Helping Your Child was developed by Cathy Creswell and Lucy Willetts from the University of Reading and University of Oxford, clinical psychologists with expertise in helping children with anxiety problems. The philosophy of the programme is the belief that parents, and carers are the experts when it comes to their child. They will have a better understanding of how their own child might respond and what will encourage and motivate them to try different things than a therapist will have.

As such, the central aim of the programme is to provide strategies for parents and carers that they can use at home to support their child for them to overcome problems with anxiety. Achieved by increasing parents' confidence in their ability to help their child overcome anxiety. As such, the philosophy of the programme is non-blaming and one that highlights positive skills and responses of parents, to build their confidence and empower them to support their children. The programme has been delivered and evaluated on an individual basis (i.e., one-to-one), and in response to demand a group programme manual that can be consistently delivered in a group format. The integration of these two foundational programmes combines EPEC's expertise in task-sharing delivery methods, reach to vulnerable and marginalised communities and wider parenting expertise with Helping your Child with Fears and Worries specialised expertise in the use of parent adjunct treatments methods for childhood anxiety.

These foundational programmes share similar theoretical foundations (of attachment, social learning and systems theory and intervention procedures (highly interactive, adult learning models, focussed skill acquisition and in vivo practice). Belsky's Multiple Determinants of Parenting (MDP) Process Model, provides the most used explanatory framework of the ecological and subjective influences on parenting and child outcomes. MDP posits that child developmental trajectories are influenced by the interaction between the child's inherent characteristics, the parenting of primary carers, the characteristics of the parent/primary care givers, the family and social environment, and wider social and economic factors. To impact on child behaviour and conduct outcomes, realistic intervention targets, based on MDP, for a psychosocial group-format parenting intervention such as EPEC include parenting, parent well-being and mental health. Family and social; encourage strategies to increase family consistency and household stability, reduce household chaos and impact of chronic stressors and social and economic such as improvements in child behaviour, parenting confidence and practices, and family functioning.

The new intervention, BAPHYC, developed from these two well-established evidence-based parenting programmes EPEC Being a Parent and Helping Your Child, is intended to provide specifically tailored parenting support to parents and other primary caregivers of children who have anxiety problems. The intervention's group-format offers the potential opportunity for participant parents and other caregivers to reduce isolation, stigma and increase social support from parents and caregivers experiencing similar problems. A peer-led, task transfer model potentially increases problem normalisation and validation, motivation for change and reduce stigma for marginalised parents and caregivers. Before undertaking a larger and costlier study it is necessary to demonstrate the viability of the novel BAPHYC intervention and associated research by testing the design and delivery of the intervention, its acceptability, and the logistics of recruitment, delivery, and data collection.

Feasibility studies are pieces of research done before a main study to answer the question "Can this study be done?" They are used to estimate important parameters that are needed to design the main study, but do not evaluate the outcome of interest; that is left to the main study.

ELIGIBILITY:
Inclusion Criteria:

* Parent/ primary caregiver, including non-biological caregiver, for index child aged 5-12 years.
* Parent-reported difficulties and concerns in managing anxiety of an index child. In households with more than one child aged 5-12 years, we ask the parents to nominate an index child whose behaviour was of greatest concern.
* Parent/ primary caregiver must have proficient written and spoken English.
* Parent/ primary must have capacity to provide informed consent to participate.

Exclusion Criteria:

Families where the parent/ parental caregiver:

* The nominated index child of the parent/ primary caregiver has a primary neurodevelopmental condition such as autism, for which parent is likely to require specialist parenting intervention.
* The parent / primary caregiver is unable to attend weekly course sessions of the BAPHYC intervention.
* The parent / primary caregiver is not living with the index child and is unlikely to have sufficient contact to implement parenting skills acquired during the BAPHYC intervention.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Parent or parental caregiver including non-biological caregiver, for index child aged 5-12 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Child Anxiety Impact Scale for Parents - change is being assessed | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  A 27-item parent-report measure assessing the impact of anxiety symptoms on the psychosocial functioning of children and adolescents (Langley, Bergman, McCracken, & Piacentini, 2004). It provides a quantitative measure of anxiety related functional impairment related to specific situations from multiple psychosocial domains (School, Social, Home/Family). It was designed as both a baseline measure and to evaluate treatment response. The respondents are asked to rate how much difficulty the child has had completing each activity due to his or her anxiety symptoms during the last month. Each item is scored on a 4-point Likert scale ("0" not at all, "1" just a little, "2" pretty much, "3" very much). Sum of subscales, or overall total score of the scale

OTHER OUTCOMES:
Treatment Acceptability Rating Scale | "immediately after the intervention/procedure/surgery"
  This 12-item self-report questionnaire (C. Day et al., 2012) uses a 4-point Likert scale to assess, (i) parenting knowledge, skills and confidence acquired (TARS KSC - 4 items yield total score 4-16) and (ii) intervention satisfaction and quality (TARS SQ - 5 items yield total score 5-20). Higher scores indicate greater acceptability and satisfaction. Three free-text items cover helpful and unhelpful participant experience
Concerns About My Child (CAMC) - Change is being assessed | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  A visual analogue scale that requires parents/caregivers to nominate, prioritise and rate up to three key concerns about their child. An idiographic measure of parental perception of child difficulties, previously used in Being a Parent trial evaluation (C. Day et al., 2012). Parents rate up to three main child emotional and behavioural concerns from 0 (not concerned at all) to 100 (could not be more concerned). Concerns were categorised into five domains: Conduct Problems, Parent-Child Relationship and Communication Difficulties, Self-Regulation, Emotional Distress and Other. The same concerns that are nominated at baseline will be re-rated at follow-up, providing a sensitive, individualised index of change
Parenting Scale (PS, 8) - Change is being assessed | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  An eight-item questionnaire that assesses dysfunctional discipline styles in parents/caregivers of children aged between 2-16 years. There are three subscales: laxness, over-reactivity and hostility. This adapted questionnaire (Kliem et al., 2018) from the Arnold O'Leary Parenting Scale assesses dysfunctional parental discipline styles yields a total score and parental verbosity, over-reactivity and laxness subscales. Lower scores indicate more positive parenting skills
Family Accommodation Scale - Anxiety (FASA) - Change is being assessed | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  This measure consists of 13 items (Lebowitz et al., 2013). The first 9 items assess the frequency of accommodations and are summed for the total accommodation score. Four additional items assess parental distress associated with accommodation (1 item), and children's short-term responses to not being accommodated (3 items). Items are rated on a 5-point scale of 0 to 4 ('Never' to 'Daily'). Total 9-item family accommodation scores range from 0 to 36, with higher scores indicating more accommodation
My Parenting Goals (MPG) - Change is being assessed | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  An idiographic measure of up to two personal parenting goals, using a visual analogue scale from 0 (could not be further from achieving my goal) to 100 (goal completely achieved), (C. Day et al., 2012)
Short Warwick Edinburgh Mental Wellbeing Scale (SWEMWBS) - Change is being assessed | "baseline, pre-intervention/procedure/surgery" and "immediately after the intervention/procedure/surgery"
  A seven-item parent wellbeing measure each rated on a 5-point Likert scale (Tennant et al., 2007). High scores represent greater mental wellbeing. SWEMWBS is sensitive to change, and the full version has been used in evaluations of parenting programmes. It had good internal consistency, α= .85. Raw SWEMWBS scores will be transformed to allow comparisons with national survey data
Goal Based Outcomes (GBO) - Changes is being assessed | "baseline, pre-intervention/procedure/surgery" and "up to nine weeks"
  This measure compares how far a person feels they have moved towards reaching a goal that they have set for themselves at the beginning of an intervention (Law, 2015.). GBOs are simply a way of deciding at the beginning of an intervention where you want to head for, and to track progress along the way, or at the end to see how far along your agreed track you have managed to get. Goal setting should occur over the first three sessions of the intervention/assessment. Each goal is given an identity number (from one to three). Once a goal is agreed, how close the respondent feels they are to reaching the goal is recorded at time one. At the end of the intervention record again how close to reaching the goal at time 2. The rating is recorded on a scale from zero to ten where 'zero' means the goal is not met in any way, 'ten' means the goal is met completely and a rating of 'five' means they are halfway to reaching the goal.

CONTACTS AND LOCATIONS:
Overall Officials: Crsipin Day, Principal Investigator — South London and Maudsley NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No
This is a feasibility study; process evalaution with a small, but targeted recrutiment sample set. We will only be looking at mechanisms of reach, engagement and delivery and completion rates. No planned detailed analysis of effect sizes will be conducted. We will share the protocol and participant information sheets.